CLINICAL TRIAL: NCT00013143
Title: Patient Profiling and Provider Feedback to Reduce Adverse Drug Events
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: SAF 99-144
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Adverse Drug Events
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Patient risk profiling (potential ADEs) w/provider feedback

INTERVENTIONS:
Behavioral: Patient risk profiling (potential ADEs) w/provider feedback

SUMMARY:
Adverse drug events (ADE) present a unique focus for error reduction. Computerized provider order entry, with embedded clinical decision support, has great promise in reducing medication errors but preventable adverse drug events may still occur despite such systems.

DETAILED DESCRIPTION:
Background:

Adverse drug events (ADE) present a unique focus for error reduction. Computerized provider order entry, with embedded clinical decision support, has great promise in reducing medication errors but preventable adverse drug events may still occur despite such systems.

Objectives:

The purpose of the study was to evaluate whether adding medication profiling (by using a retrospective drug utilization review program) to computerized provider order entry with embedded order checks (drug alerts) reduces the incidence of adverse drug events.

Methods:

Medication profiles mainly focused on possible drug-drug and drug-disease interactions, with some drug duplications. To do the medication profiles we licensed a proprietary computerized retrospective drug utilization review system. We randomly assigned over 900 patients to Usual Care or Provider Feedback. For patients in the latter group, selected providers were contacted by letter with pertinent information; electronic mail was used for follow-up contact. Clinical and other relevant data was retrospectively abstracted from the medical records for up to one year from the last medication profile for all patients. This was done by a pharmacist reviewer, using a study-derived instrument, and blinded to patient assignment. ADE incidence is the primary outcome of interest, with other outcomes such as ADE severity and preventability also assessed. We also developed and implemented provider surveys in pre- and post-profiling periods.

Status:

Pre and post survey results published. Adjunct study on clinical actions as a result of drug alerts published. Main study (profiling): manuscript in proces.

ELIGIBILITY:
Inclusion Criteria:

* patient must be alive
* patient must be currently active in GLA system
* medication for which alert was generated must be currently active
* patient provider must not be Peter Glassman

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2001-06; Study Completion 2003-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter A. Glassman, MBBS MSc, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

REFERENCES:
- [Result] Glassman PA, Belperio P, Simon B, Lanto A, Lee M. Exposure to automated drug alerts over time: effects on clinicians' knowledge and perceptions. Med Care. 2006 Mar;44(3):250-6. doi: 10.1097/01.mlr.0000199849.08389.91. PMID 16501396
- [Result] Glassman PA, Simon B, Belperio P, Lanto A. Improving recognition of drug interactions: benefits and barriers to using automated drug alerts. Med Care. 2002 Dec;40(12):1161-71. doi: 10.1097/00005650-200212000-00004. PMID 12458299
- [Result] Glassman PA, Belperio P, Lanto A, Simon B, Valuck R, Sayers J, Lee M. The utility of adding retrospective medication profiling to computerized provider order entry in an ambulatory care population. J Am Med Inform Assoc. 2007 Jul-Aug;14(4):424-31. doi: 10.1197/jamia.M2313. Epub 2007 Apr 25. PMID 17460134